CLINICAL TRIAL: NCT06366659
Title: Unraveling the Pathogenesis of Pruritus in Intrahepatic Cholestasis of Pregnancy
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2024049
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Intrahepatic Cholestasis of Pregnancy
Keywords: diagnosis; prediction; prognosis
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ICP patients: None intervention
- Healthy pregnant women: None intervention

SUMMARY:
This study hopes identify the main pruritogens of ICP pruritus and provide new insights for the diagnosis, prediction, and treatment of ICP. Details are as follows: It is planned to include ICP confirmed pregnant women and healthy pregnant women who have given birth in the Peking University Third Hospital and Sichuan University West China Second University Hospital. Then progesterone sulfate levels in plasma samples will be quantified by High Performance Liquid Chromatography-Mass Spectrometry (HPLC-MS) and itch intensity will be quantified by questionnaires. Main study endpoint: To reveal new indicators of ICP diagnosis with high accuracy: single, multiple or combined indicators of progesterone sulfates and other molecules like bile acids; Secondary study endpoint: To determine whether progesterone sulfates can be used as an early screening indicator for ICP for disease prediction, specifically whether elevated levels of progesterone sulfates predate pruritus in pregnant women with ICP.

DETAILED DESCRIPTION:
As the most common liver-related disease in pregnancy, ICP affects an average of 4% of pregnant women worldwide. In a cohort study of 12200 eligible Chinese pregnant women, the reported incidence of ICP was 6.06%. ICP is harmful to the health of both pregnant women and fetuses. For the fetus, ICP directly affects the healthy growth and smooth delivery of the fetus. Disease-related adverse events have been reported, including preterm birth, meconium contamination of amniotic fluid, fetal hypoxia, prolonged length of stay in neonatal unit, and even stillbirth. ICP has a serious impact on the physical and mental health of pregnant women, typically severe pruritus. This itching occurs mainly in the second and third trimesters of pregnancy (usually the third trimester) and tends to become progressively worse as the pregnancy progresses. It is most commonly present on the palms and soles of the feet, and some patients have generalized itching. Moreover, the itching was aggravated at night, leading to severe insomnia. Under the background of advocating multiple births in our country, the effective prevention and treatment of such diseases is particularly important.

At present, there are no effective drugs for the treatment of ICP, especially pruritus symptoms, because the molecular mechanism of ICP and its pruritus is still unclear. In this study, we have identified several endogenous potential pruritogens that can activate human MRGPRX4, the potential itch receptor of ICP pruritus, to mediate ICP pruritus based on a large number of previous cell and animal experiments. Based on clarifying the mechanism of pruritus, this project hopes to provide new biomarkers and new perspectives for the diagnosis and even prediction of the disease combined with the analysis of clinical samples. As such, health monitoring and early intervention may thus be enabled during pregnancy to benefit the treatment outcome of both the patient and child clinically. methods are as follows:

① To characterize the dynamic changes of progesterone sulfates in patients with ICP during the first, second, and third trimesters of pregnancy In cooperation with teams in the Department of Obstetrics and Gynecology of hospitals, blood samples will be collected from pregnant women at three different time points during pregnancy (including healthy pregnant women and pregnant women with ICP). A questionnaire will be completed by the pregnant women in the third trimester or by telephone follow-up after delivery. The degree of pruritus in pregnant women with ICP will be counted. The changes of progesterone sulfate levels and the degree of pruritus are characterized by the progression of pregnancy cycle. For the analysis of metabolite composition in plasma, we developed HPLC-MS based separation and quantification methods, focusing on the progesterone metabolites/derivatives of interest, including the following nine progesterone sulfates: Isopregnanolone sulfate (3β5α) (PM5S), Epipregnanolone sulfate (3β5β) (PM7S), Pregnanolone sulfate (3α5β) (PM6S), Allopregnanolone sulfate (3α5α) (PM4S), Pregnanediol sulfate (3α5β) (PM3S), Isopregnanediol sulfate (3β5α), 5β-pregnan-3α, 20α-diol-3, 20-disulfate (PM3DiS), 5α-pregnan-3α, 20α-diol-3, 20-disulfate (PM2DiS), Pregnenolone sulfate and 17-Hydroxypregnenolone sulfate. A 100 μl plasma sample is mixed with 425 μl methanol and vortexed for 10 min. After centrifugation at 14 000 g for 10 min, the supernatant is transferred to a new tube and stored at -80 ° C before HPLC-MS analysis.

② Develop diagnostic and early prediction models for ICP or pruritus symptoms. After obtaining a sufficient amount of biological samples and the metabolite analysis results, we plan to conduct effective statistical analysis and data mining based on the sample data. Using the data of related metabolites in the blood of ICP patients and healthy pregnant women in the third trimester, Receiver Operating Characteristic (ROC) curves analysis and logistic regression model will be used to find a single characteristic metabolite molecule or a combination of several metabolite molecules, which could effectively distinguish ICP patients from normal pregnant women, and serve as a new indicator with high accuracy to assist the clinical diagnosis of ICP. Furthermore, based on the analysis of blood samples in the first and second trimesters, we expect that characteristic metabolites can be mined, and the dynamic changes in their levels can even predict the probability of ICP before the onset of ICP symptoms, so as to guide the implementation of preventive measures in advance and possibly reduce the probability of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Pruritus in pregnancy
* Elevated levels of serum alanine aminotransferase (ALT) activities and total bile acids (TBA)
* Exclusion of other causes of liver dysfunction or itching

Exclusion Criteria:

* Pruritus with skin lesions such as eczema
* Pruritus of other liver-related diseases (PBC, Primary Sclerosing Cholangitis (PSC), etc.)
* Twin pregnancy
* TBA and pruritus did not relieve 4-6 weeks after delivery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants including ICP patients and healthy pregnant women without other complications will be collected form Peking University Third Hospital and Sichuan University West China Second University Hospital.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2025-08-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Progesterone metabolites (levels in plasma) | 1 year in total. Plasma samples will be collected every 3 months during the whole pregnancy of every participant. About at the last day of the month 3, month 6, and month 9 of the whole pregnancy, respectively.
  Analyze the plasma samples through HPLC-MS
Itch intensity | 1 year in total. At the last day of the month 9 of the pregnancy of participants.
  through questionnaire

SECONDARY OUTCOMES:
Total bile acids (levels in plasma) | 1 year in total. Plasma samples will be collected every 3 months during the whole pregnancy of every participant. About at the last day of the month 3, month 6, and month 9 of the whole pregnancy, respectively.
  Analyze the plasma samples through HPLC-MS

CONTACTS AND LOCATIONS:
Overall Officials: Yulong Li, Principal Investigator — Peking University
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Sichuan University West China Second University Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Privacy and research competition

REFERENCES:
- [Background] Abu-Hayyeh S, Ovadia C, Lieu T, Jensen DD, Chambers J, Dixon PH, Lovgren-Sandblom A, Bolier R, Tolenaars D, Kremer AE, Syngelaki A, Noori M, Williams D, Marin JJ, Monte MJ, Nicolaides KH, Beuers U, Oude-Elferink R, Seed PT, Chappell L, Marschall HU, Bunnett NW, Williamson C. Prognostic and mechanistic potential of progesterone sulfates in intrahepatic cholestasis of pregnancy and pruritus gravidarum. Hepatology. 2016 Apr;63(4):1287-98. doi: 10.1002/hep.28265. Epub 2015 Dec 28. PMID 26426865
- [Background] De Borre M, Che H, Yu Q, Lannoo L, De Ridder K, Vancoillie L, Dreesen P, Van Den Ackerveken M, Aerden M, Galle E, Breckpot J, Van Keirsbilck J, Gyselaers W, Devriendt K, Vermeesch JR, Van Calsteren K, Thienpont B. Cell-free DNA methylome analysis for early preeclampsia prediction. Nat Med. 2023 Sep;29(9):2206-2215. doi: 10.1038/s41591-023-02510-5. Epub 2023 Aug 28. PMID 37640858